CLINICAL TRIAL: NCT03888508
Title: Comparison of Efficacy of Sensory Integration Therapy as an Adjunct to Standard Care With Standard Care Alone in Improving Gross Motor Skills in Cerebral Palsy Children With Sensory Processing Abnormalities
Brief Title: Comparison of Efficacy of Sensory Integration Therapy in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor and Chief,Child Neurology Division,, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIT
Record Dates: First submitted 2018-05-10; First posted 2019-03-25 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Single Blind Randomized Controlled Parallel Design trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIT plus standard therapy (Experimental): Sensory interventions will include maneuvers for both hypo and hyper-reactive behaviors in five senses such as tactile, vestibular, proprioception, vision and auditory using a sensory integration kit and other items available at home Sensory integration kit will be prepared which consists of varying textures from soft to hard items (wool, jute, sand paper, velvet), picture cards, sensory brush, elastic band(Thera tube) and also usage of other home based items such as swings, sofa/bed, textured board, black board, wet chalks and paint. Each session would take approx 60 minutes/ day with each sensory stimulus given for 10-30 minutes 6 d Conventional physiotherapy, occupational,behavioural intervention and pharmacotherapy that they are already receiving as a standard therapy
  Interventions: Other: SIT
- Standard therapy alone (No Intervention): Standard therapy -Conventional physiotherapy, occupational,behavioural intervention and pharmacotherapy that they are already receiving

INTERVENTIONS:
Other: SIT — sensory integration therapy along with standard therapy.
  Primary care giver will be trained to perform sensory integration therapy at home.
  . Sensory interventions will include maneuvers for both hypo and hyper-reactive behaviors in five senses as tactile, vestibular, proprioception, vision and auditory using a sensory integration kit and other items available at home
  Daily sessions of approx 60 minutes/ day with each sensory stimulus given for 10-30 minutes 6 days in a week will be done.
  Other Names: Standard therapy
  Arms: SIT plus standard therapy

SUMMARY:
In this we are comparing efficacy of sensory integration therapy as an adjunct to standard care with standard care alone in improving gross motor skills in cerebral palsy children with sensory processing abnormalities.Existing literature points towards presence of sensory processing abnormalities in children with cerebral palsy.However, there is lack of robust evidence for usefulness of sensory integration therapy in cerebral palsy children .Standard therapy outcome in improving functional motor skills, adaptive responses are variable in children with cerebral palsy.Sensory integration therapy in addition to standard therapy may further improve adaptive and functional motor skills in children with cerebral palsy.

DETAILED DESCRIPTION:
* Study will be started after obtaining ethical clearance and registration with Clinical trials registry of India
* Hindi translation of SPCQ-2(Sensory profile caregiver questionnaire 2) by subject expert by forward and independent backward translation .
* Consecutive children of either sexes between 3-12 years with a clinical diagnosis of spastic cerebral palsy will be examined by the investigator and those having sensory abnormalities as screened by Sensory profile caregiver questionnaire 2 will be included in the study group.
* Those children who screen positive for sensory abnormalities fulfilling the inclusion criteria would be enrolled in the study after obtaining informed consent from the parents or guardian.
* Once enrolled children would be randomized into 2 groups , using a computer generated random number sequence, an interventional group receiving sensory integration therapy along with standard therapy and a group receiving standard therapy alone.
* Concealment of the random allocation would be ensured by placing the allocation sequence in serially numbered, tamper proof, opaque and sealed envelopes(by a person other than primary investigator to ensure blinding and further observation bias)
* Post - enrollment - Baseline clinical and demographic data will be recorded along with associated co morbidities (maladaptive behavior, sensory deficits and motor problems).
* Pre-intervention a baseline motor skill will be obtained using Gross Motor Function Measure -88 and behavioral assessment would be done using Child Behaviour Checklist within 7 days of starting therapy in both arms (by pediatric neurologist ,child psychologist respectively and who is unaware of the randomization and allocation to both arms to prevent observer bias).
* Pre-intervention investigator would also interact with the parents or the primary care giver and record parent's assessment of severity of sensory abnormalities in 5 main domains - auditory , visual, tactile, proprioceptive and vestibular senses on a 10 item Likert scale and also assess Quality of life using Pediatric Quality of life using Pediatric Quality of life scale
* All children would be followed at set intervals from initiation of therapy as noted below ;
* Weekly for 2 weeks then fortnightly for next 10 weeks to ensure proper technique and compliance.
* At 3 months the blinded outcome assessor and child psychologist will re evaluate the enrolled candidate to determine for any change by using Gross Motor Function Measure -88 , 10 item parent rated Likert scale, Child Behaviour Checklist and Pediatric Quality of life as compared to baseline within 7 days of completion of therapy in both arms

The first visit would be primarily aimed at reinforcing the techniques of therapy and clarifying parent's doubts. At 3 month visit child would be evaluated and re-assessed using the scores- 10 item Likert scale rated by parents, Gross Motor Function Measure -88 and Pediatric Quality of life scale . Parents would be encouraged to bring one random home video of child doing activity-based therapy at 2 weeks wherever feasible . The video would be used for ,

* Assessing the correct technique
* Suggesting modifications in the activity schedule if required
* Helps in ensuring adherence to technique

Compliance would be ensured by the

* Activity log
* Telephonic re-enforcement from the primary investigator weekly

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex aged 3 to 12 years clinically diagnosed to have spastic cerebral palsy

  * Definite Sensory processing abnormality defined as (more than 2 standard deviations below the mean) in at least one of the nine domains of sensory profile -2 questionnaires
  * GMFCS either I, II or III
  * Minimum visual acuity of 6/60
  * IQ/SQ>70.
  * Either parent should be willing to come for follow up.
  * Stable pharmacotherapy, conventional physiotherapy, behavioral interventional therapy and occupational therapy for last 4 weeks

Exclusion Criteria:

* Receiving /received Sensory Integration therapy in the past 6 months
* Hemi paretic and mixed cerebral palsy
* Children of either sex aged 3 to 12 years clinically diagnosed to have spastic cerebral palsy

  * Fixed contractures and deformities in lower limbs affecting stance and gait.
  * Received botulinum toxin injection or undergone orthopedic corrective surgery in the past one year prior to enrolment
  * Refractory epilepsy as per ILAE definition.
* Failure of adequate trials of two tolerated, appropriately chosen and used antiepileptic drug schedules (whether as mono therapies or in combination) to achieve sustained seizure freedom

  * Autistic features, Attention Deficit Hyperactivity Disorder, Specific Learning Disability satisfying Diagnostic and Statisitical Manual of Mental disorders V criteria for these disorders
  * Current clinically significant medical disorders (as determined by Investigator)
* Cardiovascular (e.g. Congestive Cardiac Failure)
* Respiratory (e.g. severe asthma, severe pneumonia)
* Gastrointestinal (e.g. upper GI bleed)
* Renal (e.g. acute renal failure )
* Hepatic (e.g. acute liver failure)
* Hematologic or other medical disorders

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Mean change in GMFM-88 Score from baseline | 3 months
  Gross Motor Function Measure (GMFM-88)
  The gross motor function measure-88 (GMFM-88) is a well-known scoring system, which assesses gross motor development in children with CP over time in 5 domains
  A (lying and rolling), 17 items
  B (sitting), 20 items
  C (crawling and kneeling), 14 items
  D (standing), 13 items;
  E (walking, running, and jumping), 24 items.

SECONDARY OUTCOMES:
Mean T score change from baseline in CBCL | 3 months
  Child behaviour checklist (CBCL)-140 items-Self-administered or administered through an interview; norm referenced comprehensive measure of behavior; examines aggression, hyperactivity, bullying, conduct problems, defiance, violence Three formats: Teacher Report Forms, Youth Self-Reports, and Direct Observation Forms Yields standard scores: Total Competence, Total Problems, Internalizing, Externalizing, Attention Problems
Mean score change from baseline in Pediatric quality of life scale from baseline | 3 months
  PedsQL-The PedsQL measurement model is a modular approach to measure health related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. The PedsQL measurement model integrates seamlessly both generic core scales and disease-specific modules into one measurement system. It's a brief 23 item multi-dimensional scale, comprising questions in physical, emotional, social and school functioning sectors. Takes around 4 minutes to administer the scale. Has both self-report and proxy report for the children for various age groups (ages 2-18; Child Self-Report Ages 5-7, 8-12, 13-18; Parent Proxy-Report Ages 2-4, 5-7, 8-12, 13-18yrs ). It was found to be reliable between raters and across time.
Mean score change from baseline in parent rated 10 item Likert scale | 3 months
  Likert scale-This is a scale designed to assess the severity of sensory abnormalities in children as per parents. Around 10 questions have been used, 2 each from -visual, tactile, vestibular, proprioceptive and auditory domains. These questions have been framed based on the most common sensory symptoms observed in these children. The scale rates from 1 to 5 , where 1 indicates the lower end of symptom spectrum and 5 the highest end. It is used pre as well as post intervention to compare for any change in sensory processing abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, M.D, Principal Investigator — Professor
Locations (1):
- All india institute of Medical sciences, Delhi, South Delhi, India

IPD SHARING:
Plan to Share IPD: No